CLINICAL TRIAL: NCT01190722
Title: A Randomized Study Comparing Etoricoxib and Diclofenac Sodium in Post Hallux Valgus Surgery Pain
Brief Title: A Study Comparing Etoricoxib and Diclofenac Sodium in Post Hallux Valgus Surgery Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study site was closed down
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jan Jakobsson, Adj. Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201001HV
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Hallux Valgus; Postoperative Pain
Keywords: Day case surgery; postoperative pain; NSAIDs; Coxibs
MeSH Terms: conditions — Hallux Valgus; Pain, Postoperative | interventions — Etoricoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- etoricoxib (Experimental): active study drug, coxib
  Interventions: Drug: etoricoxib
- diclofenac (Active Comparator): active traditional NSAID control
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: etoricoxib — 120 mg once daily for the 1st 6 postoperative days
  Arms: etoricoxib
Drug: Diclofenac — 50 mg oral 3 times daily the 1st 6 postoperative days
  Arms: diclofenac

SUMMARY:
The investigators hypothesize that cyclooxygenas-II-selective inhibitors (Coxibs) provide a better patients assessed overall satisfaction when used for pain management after elective hallux valgus surgery as compared to traditional Non-steroidal anti-inflammatory drugs (NSAIDs).

DETAILED DESCRIPTION:
The aim of the present study is to compare patients' satisfaction with pain medication during the first 7 first postoperative days following elective hallux valgus surgery in general anaesthesia between etoricoxib and diclofenac in a prospective randomised double-blind study design.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physiological class 1-2 patients
* aged 18-65 years
* scheduled for elective hallux valgus surgery in general anesthesia

Exclusion Criteria:

* NSAID allergy
* liver disease
* renal disease
* uncontrolled cardiovascular disease
* Lithium therapy
* chronic pain
* regular analgesia use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11-10 (Actual); Primary Completion 2010-12-11 (Actual); Study Completion 2010-12-12 (Actual)

PRIMARY OUTCOMES:
Patients Global Evaluation of Study Medication | postoperative day 1-6
  Patients self-assessment of global satisfaction with pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jakobsson, Professor, Principal Investigator — Karolinska Institutet